CLINICAL TRIAL: NCT04805762
Title: Your COACH Next Door Study. Dutch Title: Your COACH Next Door Studie.
Brief Title: Your COACH Next Door Study
Acronym: YCND
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1292
Record Dates: First submitted 2021-03-11; First posted 2021-03-18 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with overweight or obesity following the lifestyle intervention YCND: Children with overweight or obesity that are participant of the lifestyle intervention YCND
  Interventions: Other: Your COACH Next Door

INTERVENTIONS:
Other: Your COACH Next Door — Children in the study are attending the lifestyle intervention Your COACH Next Door. A coach is supporting the child and it's family to reach their goals regarding lifestyle.

SUMMARY:
Your COACH Next Door (YCND) is a lifestyle intervention connecting children with overweight and their families with a coach close to home.

This study goal is to examine the effects of YCND for children and their families, (on their health, quality of life), and a process evaluation (process of the lifestyle intervention, and satisfaction for children, families and healthcare givers)

DETAILED DESCRIPTION:
Childhood overweight and obesity in an increasing problem worldwide. Among other, childhood obesity is associated with type 2 diabetes, cardiovascular disease, NAFLD and decreased quality of life. In 2016 the lifestyle intervention Your COACH Next Door (YCND) was founded in Maastricht, The Netherlands, as a tailored, network approach for children with overweight and obesity. YCND is following the example of COACH, the tailored lifestyleintervention for childhood obesity of the expertise centre of the MUMC+ hospital.

YCND is connecting children with overweight and their families with a coach close to home.

This study goal is to examine the effects of YCND for children and their families, (on their health, quality of life), and a process evaluation (process of the lifestyle intervention, and satisfaction for children, families and healthcare givers)

ELIGIBILITY:
Inclusion Criteria:

* Participant of the YCND lifestyle intervention.
* Having overweight or obesity
* Younger than 18 years at inclusion

Exclusion Criteria:

* No exclusion criteria

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with overweight or obesity, participant of the Your COACH Next Door lifestyleintervention.
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Weight | Every consult, primary outcome at 1 year, 2 years and 3 years of intervention.
  Weight measured as change in BMI z-score

SECONDARY OUTCOMES:
Presence of comorbidities | Measured at baseline and yearly until 3 years after start of intervention.
  Presence of comorbidities measured in questionnaires, in which families and healthcare professionals can indicate if the child suffers from comorbidities (insulin resistance, DM II, hypertension, NAFLD, cardiovascular diseases) occur in the child.
QOL (quality of life) | Measured at baseline and yearly until 3 years after start of intervention.
  Quality of life as measured with a validated questionaire
Healthy eating pattern | Measured at baseline and yearly until 3 years after start of intervention.
  Healthy eating pattern of the child as measured with a questionnaire (combination of Dutch Guidelines for healthy eating for children), to determ if the child is eating healthier or less healthy after start of the intervention.
Physical activity behaviour | Measured at baseline and yearly until 3 years after start of intervention.
  Physical activity behaviour of the child as measured with a validated questionnaire for children.
Patient satisfaction | Measured at baseline and yearly until 3 years after start of intervention.
  Patient satisfaction regarding the YCND-program measured with a combination of a questionnaire and an interview.
Healthcare giver satisfaction | Measured at baseline and yearly until 3 years after start of intervention.
  Healthcare giver satisfaction regarding the YCND-program measured with a questionnaire and an interview.
Process evalution | Measured at baseline and yearly until 3 years after start of intervention.
  Process evalution, primarily measured as consultations visited by the child

CONTACTS AND LOCATIONS:
Overall Officials: Anita CE Vreugdenhil, Dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided